CLINICAL TRIAL: NCT01331044
Title: Efficacy and Acceptability of Ready to Use Therapeutic Food (RUTF) in Children Aged 6-24 Months With Severe Acute Malnutrition in Bangladesh
Brief Title: Ready to Use Therapeutic Food (RUTF) in Severe Malnourished Children
Acronym: RUTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: International Atomic Energy Agency (Other Government); Washington University School of Medicine (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-09023
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-06

CONDITIONS: Severe Acute Malnutrition
Keywords: RUTF; Severe Acute Malnutrition; Children; Body composition; Microbiota; Short Chain Fatty Acid; Acceptability of RUTF; Edema free 15 percent weight gain; Changes in body composition; Gut microbiota; Genome wide association
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RUTF (Experimental): Ready to use Therapeutic Food (RUTF) Plumpy nut.
  Interventions: Dietary Supplement: Plumpy Nut
- Khichuri - Halwa (Active Comparator): Cereal Legume
  Interventions: Dietary Supplement: Khichuri and Halwa

INTERVENTIONS:
Dietary Supplement: Plumpy Nut — to RUTF will receive commercially available RUTF (Plumpy nut) in a total of 200 kcal/kg.day in a sequential manner (Plumpy nut will be offered ~ 125 kcal/kg in 1st 24 hours, ~ 150 kcal/kg in 2nd 24 hours, then~200k cal/kg by the third day).
  Arms: RUTF
Dietary Supplement: Khichuri and Halwa — Day 1: Milk suji, 10ml/kg/ feed for 11 feed & halwa 10gm/kg; 2 feed per day 125kcal/kg.day
  Day 2: Milk suji, 10ml/kg/ feed for 11 feed & halwa 10gm/kg; 2 feed per day & khichuri 10gm/kg; 2 feed per day 150kcal/kg.day
  Day 3: Milk suji 100, 10ml/kg/ feed for 11 feed & halwa 10gm/kg; 2 feed per day & khichuri 10gm/kg; 2 feed per day 175kcal/kg.day
  Day 4: Milk suji 100, 10ml/kg/ feed for 11 feed & halwa 10gm/kg; 3 feed per day & khichuri 10gm/kg; 3 feed per day 200kcal/kg.day
  Day 5 onward: Milk suji 100, 10ml/kg/ feed 6 hourly (4 feed per day) & halwa 20gm/kg; 3 feed per day & khichuri 20gm/kg; 3 feed per day 200kcal/kg.day
  Arms: Khichuri - Halwa

SUMMARY:
1. RUTF would be more effective (quicker catch-up growth by promoting more tissue accrue resulting decrease stay in rehabilitation ward) in treating children with SAM during the rehabilitation phase than khichuri /halwa;
2. RUTF would be acceptable to the children and their mothers/caregivers;
3. Malnutrition is not caused solely by lack of food, but also by impaired utilization of the food that is ingested. The ability of the gut to absorb nutrients from the diet is associated with the host's 'human' genotype, the host's gut microbiota and its gene content (the microbiome).

DETAILED DESCRIPTION:
We propose to conduct a research study to compare the acceptability and efficacy of RUTF with that of the cereal-based diets in the management of hospitalised SAM children in Bangladesh. After completion of the initial acute phase treatment (for diarrhoea, lower respiratory tract infection/pneumonia, severe anaemia, fever, sepsis, electrolyte imbalance, and/or anorexia) in the Longer Stay Ward/ Special Care Ward of the Dhaka Hospital, the children will be transferred to the NRW according to the enrolment criteria. Once the children fulfil all the criteria for entry into the study and written consent to their participation is obtained from respective parents/guardian, they will be randomly allocated to: (i) the standard cereal-based foods, namely khichuri and halwa, or (ii) RUTF. Randomization will be done according to computer-generated random numbers using permuted blocks with block lengths of four and six. For understandable reasons, the dietary therapy can't be blinded. The assigned treatment packages will be kept in closed opaque envelopes until the same serial number is assigned to an enrolled child. Participating children will be discharged from NRW according to the new WHO growth standard (WHO, 2009), which explicit , at least after seven days stay completed there or until achieving a weight gain of 15% , for non-oedematous child. On the other hand for oedematous child after oedema free if WHZ is ≥-3; however if oedema free WHZ is <- 3 then the child will be discharge after achieving 15% weight gain. In both the groups, the acceptability of the allocated diet, both by the children and their respective mothers/caregivers, the rate of weight gain and anthropometric measurements, and adverse event will be systematically recorded for analyses. Khichuri/halwa group will be given diet as per standardized management protocol of NRW of the Dhaka Hospital. On the other hand, children allocated to RUTF will receive commercially available RUTF (Plumpy nut) in a total of 200 kcal/kg.day in a sequential manner (Plumpy nut will be offered ~ 125 kcal/kg in 1st 24 hours, ~ 150 kcal/kg in 2nd 24 hours, then~200k cal/kg by the third day). We will also examine if the weight gain of the children is associated with increase in the lean body mass or in the body fat mass by assessing their body composition, Changes in body composition after dietary intervention in SAM children will be assessed by non-invasive technique using stable isotope tracer (deuterium oxide). For this, after collection of baseline urine and saliva samples a known quantity (5 gm) of deuterium oxide labelled water will be given to all study children. Enrichment of deuterium in body water will be measured to estimate total body water (TBW). Enrichment reaches a plateau after 3-5 hours. According to the recommendation from International Atomic Energy Agency (IAEA) field manual, two post-dose saliva samples will be collected at 3rd and 4th hours. The concentrations of deuterium in saliva samples will be measured with Fourier Transform Infrared Spectrometer (FTIR). The urine specimens will be analyzed using Isotope Ratio Mass Spectrometry (IRMS). From measured TBW we would estimate the fat free mass (FFM). Body fat mass (FM) is the difference between body weight and fat free mass. This procedure will be repeated in same sequence in all study children at the end of dietary intervention when the study child achieve discharge criteria. In addition to the above mentioned procedures, anthropometric measures such as mid-arm circumference, triceps skin fold thickness, arm fat area and arm muscle area would also be routinely recorded along with other morbidity data.

We wish to leverage the ongoing scientific collaboration among University of Virginia, Center for Genome Sciences at Washington University School of Medicine, USA and ICDDR,B to gain insight into the influence of human genetic polymorphisms and gut microbiome on malnutrition, in order to provide a foundation for new treatment and prevention programs on a population-wide basis.

ELIGIBILITY:
Inclusion Criteria:

1. Children with SAM, defined as WH <- 3 Z score of WHO standard and/or bipedal nutritional oedema (according to WHO growth standard)
2. Sex: Either
3. Age: 6-24 months
4. Completed acute (stabilization) phase management and regaining appetite
5. No signs of concurrent infection (e.g. diarrhoea, lower respiratory tract infection/pneumonia, severe anaemia, fever, sepsis, electrolyte imbalance, etc.)
6. Mothers/caregivers agreed to stay in the NRW until child achieve desired discharged criteria.
7. Informed consent given by the parent or guardian.

Exclusion Criteria:

1. Children without fixed residential address
2. Children with tuberculosis or any congenital/acquired disorder
3. Any physical condition that affects normal feeding of the children e.g. Cleft lip or palate.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2009-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of weight gain | 14 days
  During stay in nutrition rehabilitation unit, Dhaka Hospital

SECONDARY OUTCOMES:
Days require to achieve oedema free discharge criteria and other anthropometric changes | 14 days
  Weight for length -2 SD or 15 percent weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Sayeeda Huq, MBBS, MIPH, Principal Investigator — International Centre for Diarrhoea Diseases Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Bangladesh, Dhaka, Bangladesh